CLINICAL TRIAL: NCT00138372
Title: Human Immunity to MSP-1 in Western Kenya
Status: Completed | Type: Observational
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, James Kazura, Distinguished University Professor School of Medicine, Case Western Reserve University
Other Study IDs: 04-110
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: malaria; immunity; MSP-1; Kenya; infants
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Adult Repeat Cross-Sectional study (ARCS): This group will be enrolled from the sub-location of Kanyawegi, Kisumu District, Nyanza Province.
- Prospective Infant Cohort study (PIC): will be a clinic-based study recruiting infants attending Chulaimbo Rural Health Training Center (CRHTC), Maseno Division, Kisumu District, Nyanza Province for routine immunizations.
- Normal volunteers: will be recruited from the CWRU/UHCMC area as well as general local community.

SUMMARY:
This is a study of 125 healthy male and female Kenyan adults aged 18 years and above, and 300 healthy male and female Kenyan infants enrolled at 1 month of age and followed to 3 years of age. Twenty healthy adults (US residents) who have no self-reported history of Malaria exposure, infection or travel to malaria endemic areas of the world will serve as Malaria Naive Negative Controls. The proposed study represents a continuation of molecular and immunologic studies done in human populations describing mechanisms of protection against malaria infection and disease. Human investigation of those experiencing natural exposure to malaria infections are justified since they will eventually be the target population for testing malaria vaccine safety and efficacy.

DETAILED DESCRIPTION:
This study will include two major populations: (1) the Adult Repeat Cross Sectional study (ARCS) will involve 125 healthy Kenya-residents male and female aged 18 years and above; and (2) the Pediatric Infant Cohort (PIC) will include 300 healthy male and female infants who are residents of Kenya. In addition, 20 healthy adult US residents, who have no self-reported history of malaria exposure, infection or travel to malaria endemic areas of the world, will serve as Malaria Naive Negative Controls (MNNC). The adult (ARCS) study will consist of 6 venous blood donations to be completed in one year. The primary outcome of the ACRS is to determine the stability of Immune responses to MSP-1 who are clinically protected against P. falciparum infections and the secondary outcome is to measure the level and stability of MSP-1 specific IIA activity, MSP-1 specific T-cell memory phenotypes and immune functions and lastly, to determine the MSP-1 genotypes. The PIC study is both home and clinic-based. The overall duration of this study will be three years. The subjects will be recruited during their routine immunizations visit. The data and sample collections consist of monthly home-visits interspersed by clinic-visits every 6 months until the child reaches 3 years old. The primary outcome of the PIC study is to evaluate the development of humoral and cellular immunity to MSP-1 in healthy children in relation to their history of P. falciparum infections, number of episodes of uncomplicated acute malarial infections in the first 3 years of life and secondary outcome is to measure the acquisition of MSP-1 specific IIA activity, shifts in T-cell memory phenotypes and amalaira-specific immunity and their association with the history of exposure to P. falciparum MSP-1 alleleic variants. For the MNNS study, the primary objective is to optimize molecular and immunologic assays to be used in Kenya and to determine background level responses in healthy adult and the secondary outcomes aims to measure the level of MSP-1 specific IIA-activity, T-cell memory phenotypes and any non-specific immunity to malaria antigens and to provide negative control DNA for P. falciparum detection and genotyping studies. The result of these studies will provide insight into how the frequency and intensity of prior malaria infection and antigenic polymorphism influence the generation and maintenance of T-cell memory and AB responses to merozoite surface proteins in humans.

ELIGIBILITY:
Inclusion Criteria:

1. Permanent residency in the study area for ARCS study and within 50 km of Chulaimbo Rural Health Training Center for PIC study.
2. Healthy by medical examination.
3. Understood and signed written informed consent and is willing to participate in the study.
4. ARCs study participants must be older than 18 years of age, and PIC study participants will be enrolled at 1 month and followed until 3 years of age.
5. Study participant willing to attend scheduled follow up visits at clinic and willing to have field assistant make home visits during follow-up.

Exclusion Criteria:

1. Hemoglobin <5 g/dl for children, <10 g/dl for adults.
2. Received a blood transfusion within the past 6 months for adults or ever for children.
3. Presence or signs of severe complicated falciparum malaria (WHO, 1989).
4. Women who are self-reported to be pregnant.
5. Unwilling or unable to continue participation.

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population will consist of 125 healthy male and female adults older than 18 years from a rural area of Western Kenya AND 300 healthy male and female infants from Western Kenya enrolled at 1 month of age and followed until the age of 3 years.
  Normal volunteers will be recruited from the CWRU/UHCMC area as well as general local community.
Sampling Method: Non-Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2004-07; Primary Completion 2008-09 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James W Kazura, M.D., Principal Investigator — Case Western Reserve University
Locations (1):
- Kenya Medical Research Institute, Kisumu, Kenya